CLINICAL TRIAL: NCT04696731
Title: A Phase 1A/1B Multicenter Study Evaluating the Safety and Efficacy of ALLO-316 With Cyclophosphamide/Fludarabine Lymphodepletion Alone or Including ALLO-647 in Subjects With Advanced or Metastatic Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: Safety and Efficacy of ALLO-316 in Subjects With Advanced or Metastatic Clear Cell Renal Cell Carcinoma
Acronym: TRAVERSE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-316-101
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced/Metastatic Clear Cell Renal Cell Carcinoma
Keywords: CAR T; Cell Therapy; Allogeneic Cell Therapy; Cellular Immuno-therapy; AlloCAR T; ALLO-316; ALLO-647; CCRCC; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALLO-647, ALLO-316 (Experimental)
  Interventions: Genetic: ALLO-316; Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ALLO-316 — ALLO-316 is an allogeneic CAR T cell therapy targeting CD70
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion

SUMMARY:
This is a Phase 1 dose escalation study following a 3+3 study design. The purpose of the TRAVERSE study is to assess the safety, efficacy, and cell kinetics of ALLO-316 in adults with advanced or metastatic clear cell renal cell carcinoma after a lymphodepletion regimen comprising fludarabine, cyclophosphamide, with or without ALLO-647 to define a Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma with a predominant clear cell component.
* Must have received a checkpoint inhibitor and a VEGF inhibitor in the advanced and/or metastatic setting.
* At least one measurable lesion as defined by RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Absence of donor (product)-specific anti-HLA antibodies (DSA).
* Adequate hematological, renal, liver, pulmonary, and cardiac functions.

Exclusion Criteria:

* Central nervous system (CNS) metastatic disease (unless controlled and stable for at least 4 weeks), leptomeningeal disease, or cord compression.
* Clinically significant CNS dysfunction.
* Any other active malignancy within 3 years prior to enrollment.
* Prior treatment with anti-CD70 therapies.
* Current thyroid disorder (including hyperthyroidism) with the exception of hypothyroidism controlled on stable dose of hormone replacement therapy.
* Prior treatment with anti-CD52 monoclonal antibody in the past 12 months.
* Patients unwilling to participate in the extended safety monitoring period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects experiencing Dose Limiting Toxicities at increasing doses of ALLO-316 | 28 days
Proportion of patients experiencing Dose Limiting Toxicity with ALLO-647 in combination with fludarabine/cyclophosphamide administered prior to ALLO-316 | 33 days

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Namdari H, Rezaei F, Heidarnejad F, Yaghoubzad-Maleki M, Karamigolbaghi M. Immunoinformatics Approach to Design a Chimeric CD70-Peptide Vaccine against Renal Cell Carcinoma. J Immunol Res. 2024 Jan 27;2024:2875635. doi: 10.1155/2024/2875635. eCollection 2024. PMID 38314087
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350